CLINICAL TRIAL: NCT06685887
Title: Phase Ⅱ Study of Systemic Chemotherapy and Immune Checkpoint Inhibitors Combined With Hyperthermic Intraperitoneal Chemotherapy in the Treatment of Gastric Cancer Patients With Peritoneal Metastasis
Brief Title: A Clinical Study Evaluating the Efficacy of Systemic Chemotherapy and Immune Checkpoint Inhibitors Combined With Hyperthermic Intraperitoneal Chemotherapy in the Treatment of Gastric Cancer Patients With Peritoneal Metastasis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Collaborators: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UHCT230584
Record Dates: First submitted 2024-06-30; First posted 2024-11-13 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2024-06

CONDITIONS: Gastric Cancer
Keywords: Peritoneal Metastasis; HIPEC; SOX; Tislelizumab
MeSH Terms: conditions — Stomach Neoplasms | interventions — Hyperthermic Intraperitoneal Chemotherapy; Immune Checkpoint Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HIPEC combined with SOX and Tislelizumab (Experimental): The participants volunteering to take HIPEC combined with SOX and immune checkpoint inhibitors will be assigned to this group.
  Interventions: Drug: HIPEC; Drug: SOX; Drug: Immune Checkpoint Inhibitors

INTERVENTIONS:
Drug: HIPEC — HIPEC treatment (Oxaliplatin, physiological saline at 43°C for 60 min) was performed after the Laparoscopic exploratory surgery.
Drug: SOX — Oxaliplatin, 130 mg, i.v. + S-1 (40 mg per dose for BSA <1.25; 60 mg per dose for BSA 1.25 to 1.5; 60 mg per dose for BSA ≥1.5, twice daily for each treatment cycle d1-14, q3w
Drug: Immune Checkpoint Inhibitors — Tislelizumab, 200 mg, q3w

SUMMARY:
This study is a single-center, prospective, phase II clinical trial aimed at assessing the impact of HIPEC combined with systemic chemotherapy and immune checkpoint inhibitors on the R0 resection rate in patients with peritoneal metastasis from gastric cancer. Furthermore, it seeks to analyze the effects of this treatment strategy on overall survival (OS), progression-free survival (PFS), PCI and adverse reaction rates.

DETAILED DESCRIPTION:
Gastric cancer with peritoneal metastasis represents an advanced stage of the disease, with a very poor prognosis for patients. It is crucial to develop more effective treatment options to improve their prognosis. CRS with HIPEC has shown promise in extending survival for these patients. Currently, a PCI value ≥12 is widely recognized as significantly impacting the prognosis of gastric cancer peritoneal metastasis.

Recent clinical trials have resulted in the global endorsement of immune checkpoint inhibitors as a third-line therapy for gastric cancer. In March 2020, the National Medical Products Administration (NMPA) granted approval for nivolumab to be used in advanced or recurrent patients with gastric or esophagogastric junction adenocarcinoma who have received two or more systemic treatments.

However, there remains a lack of widely accepted effective treatment regimens for patients with peritoneal metastasis of gastric cancer. The CSCO recommends that such patients be referred for standard advanced gastric cancer treatments or consider participation in clinical trials. Consequently, our center has developed a comprehensive treatment protocol involving systemic chemotherapy (SOX), immune checkpoint inhibitors (Tislelizumab) and HIPEC, aiming to investigate the safety of this regimen and further enhance the prognosis of patients with peritoneal metastasis from gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

1. 18-75 years
2. Men, or non-pregnant and non-lactating women
3. Pathological diagnosis as gastric malignant tumor
4. diagnosis of peritoneal metastasis [peritoneal cancer index (PCI) ≤ 12 points] by laparoscopic exploration
5. Normal major organ function:

1) HB ≥ 90 g/L； ANC ≥ 1.5×109/L; plt ≥125×109/L; 2) TBIL<1.5ULN; ALT, AST <2.5ULN; Cr≤1.25ULN; ALB ≥ 30 g/L 6. Not receive radiation therapy, chemotherapy, targeted therapy, or immunotherapy.

7. Eastern Cooperative Oncology Group Performance Status (ECOG): 0-1 8. Patients are volunteers, have signed informed consent, and agree to cooperate with investigators in data collection.

Exclusion Criteria:

1. Patients have other malignant tumors within the past 5 years.
2. Patients use immunosuppressant within 30 days prior to the initial use of tirelizumab, excluding nasal sprays and physiological doses of inhaled corticosteroids or systemic steroids from consideration.
3. Patients have a documented history of ongoing autoimmune conditions or prior autoimmune diseases.
4. Patients are allergic to oxaliplatin, S-1, other related chemotherapy drugs or immune checkpoint inhibitors.
5. Patients with epilepsy or other mental disorders.
6. Patients who are unable to undergo surgery due to severe heart, lung and vascular diseases.
7. Pregnant or lactating women.
8. Patients with other distant metastasis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-02-15 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
R0 resection rate | 1 year
  The proportion of patients who achieved R0 resection

SECONDARY OUTCOMES:
1,2,3-year OS rate | up to 12/24/36-months follow-up
  The proportion of patients who will be alive within 1/2/3 years after receiving surgery
Progression-free Survival | up to 36-months follow-up
  Percentage of all patients who did not experience disease progression or death.
Incidence and severity of adverse reactions and serious adverse events | up to 36-months follow-up
  The incidence of adverse events and serious adverse events (referring to CTCAE 5.0) will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Kaixiong Tao, PhD, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Wuhan Union Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No